CLINICAL TRIAL: NCT07355062
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Veverimer in Adults With CKD and Metabolic Acidosis (The REVIVE Study)
Brief Title: A Study to Evaluate the Efficacy and Safety of Veverimer for the Treatment of Metabolic Acidosis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Renibus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REN-012
Record Dates: First submitted 2025-11-25; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: CKD; Metabolic Acidosis
Keywords: CKD; Metabolic Acidosis; Veverimer; STS5; Bicarbonate
MeSH Terms: conditions — Acidosis | interventions — veverimer

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 2:1 to veverimer or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Veverimer (Experimental)
  Interventions: Drug: Veverimer
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Veverimer — Group 1: 9 g veverimer BID
  Arms: Veverimer
Drug: Placebo — Group 2: 9 g PBO BID
  Arms: Placebo

SUMMARY:
The purpose of this 26 week study is is to evaluate the efficacy and safety of veverimer in treating adults with moderate-to-severe chronic kidney disease (CKD) and metabolic acidosis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* ≥ 18 years old (male/female)).
* CKD with eGFR < 60 mL/min/1.73m²; not expected to need dialysis/ transplant during study.
* 2 SBC values 12-21 mmol/L within 6 months pre-screening
* During screening: 2 central SBC values 12-21 mmol/L
* Willing to maintain stable diet .
* Expect to keep oral alkali therapy dose stable.
* Women of childbearing potential: negative pregnancy test and agree to abstinence or contraception.

Exclusion Criteria:

* Any participant deemed by the Investigator to be an inappropriate candidate for physical performance testing (e.g., severe musculoskeletal pain, non-ambulatory status) or with a screening STS5 time < 10 seconds (i.e., very mobile).
* Any participant deemed by the Investigator to be an inappropriate candidate for CPET (e.g., advanced chronic obstructive pulmonary disease [COPD], major cardiovascular [CV] event in last 6 months, systolic blood pressure [SBP] > 200 mmHg or diastolic blood pressure [DBP] > 120 mmHg). Only applicable to sites performing CPET and if the participant will take part in CPET.
* History or current diagnosis of:

  1. Clinically significant gastroparesis or a history of bariatric surgery.
  2. Bowel obstruction, swallowing disorders, severe gastrointestinal disorders, including inflammatory bowel disease, major gastrointestinal surgery, or known active gastric/duodenal ulcers.
  3. Severe recurrent diarrhea or severe recurrent constipation, in the opinion of the Investigator.
  4. Pernicious anemia, atrophic or autoimmune gastritis, achlorhydria or hypochlorhydria.
* Active Helicobacter pylori infection at screening.
* Active, recurrent, or metastatic malignancy at the start of screening.
* History of malignancy, except under the following conditions:

  1. Carcinoma in situ (e.g., of the cervix, breast, or bladder) that has been completely excised and shows no evidence of residual disease.
  2. Non-melanoma skin cancers (e.g., basal cell carcinoma, squamous cell carcinoma) that have been completely excised and show no evidence of recurrence.
  3. Low grade prostate cancer, in the opinion of the Investigator (i.e., no metastasis, Gleason score < 6), with no significant worsening for > 6 months prior to the screening visit.
  4. Any other malignancy that was treated with curative intent and has been in complete remission for ≥ 5 years prior to the screening visit.
* Evidence of acute fluid overload or history of recurrent fluid overload, in the opinion of the Investigator.
* Screening hemoglobin < 10 g/dL.
* Presence of primary respiratory alkalosis, as assessed by venous blood gas (VBG) analysis at time of screening.
* Serum gastrin level > 500 pg/mL.
* Investigational medication administration within 28 days prior to start of screening.
* Use of GI polymer binders or sodium zirconium cyclosilicate within 28 days prior to the start of screening or have an expectation to initiate treatment during the study.
* Use of acid reducing drugs, including potassium competitive acid blockers, H2-blockers or PPIs within 28 days prior to the start of screening or have an expectation to initiate treatment during the study.
* Use of GLP-1 inhibitors within 6 months prior to the start of screening or have an expectation to initiate treatment during the study.
* Participants that are taking any of the following medications and have not been on a stable dose for at least 28 days prior to screening or have an expectation to change dose during the study: diuretics, non-ophthalmic carbonic anhydrase inhibitors, diabetes drugs, RAAS inhibitors, calcium or magnesium supplements, non polymer phosphate binders, and SGLT-2 inhibitors. These medications also should not be started during the study.
* Participants that are taking more than 30 units of insulin daily.
* History of alcoholism or drug/chemical abuse within 1 year prior to the start of screening, in the opinion of the Investigator.
* Current, regular use of inhaled/ingested cannabis/THC products.
* Inability to take the IP or otherwise comply with the protocol.
* Any medical condition, uncontrolled systemic disease or serious concurrent illness that would significantly decrease study compliance or jeopardize the safety of the participant or affect the validity of the trial results, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Veverimer by measuring change in serum bicarbonate concentration (SBC) | Visits: Screening to Day 168
Efficacy of Veverimer in improving physical performance as assessed by the Sit-to-Stand 5 times test (STS5). | Visits: Screening to Day 168

SECONDARY OUTCOMES:
Efficacy of Veverimer in improving physical performance as assessed by the the 6-minute walk test (6MWT). | Visits: Screening to Day 168
Change in Kidney Disease Quality of Life Physical Function Domain (KDQOL-PFD) | Visits: Screening to Day 168
  Patients answer the following 10 questions with: "Yes, limited a lot (0 points)"; "Yes, limited a little (5 points)"; or "No, not limited at all (10 points)"
  * Vigorous activities, such as running, lifting heavy objects, participating in strenuous sports
  * Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf
  * Lifting or carrying groceries
  * Climbing several flights of stairs
  * Climbing one flight of stairs
  * Bending, kneeling, or stooping
  * Walking more than a mile
  * Walking several blocks
  * Walking one block
  * Bathing or dressing yourself Score can range from 0-100, with a higher score being a better outcome.
Improvement in Patient Global Impressions Scale - Severity (PGI-S) | Visits: Screening to Day 168
  Patients answer 1 question throughout the duration of the study: How would you rate your current level of physical functioning (mobility and ability to do every day physical activities)? Poor, Fair, Good, Very good, Excellent. Score can be 1-5, with a higher score being a better outcome.
Change in peak VO2 (peak volume of oxygen) in participants undergoing CPET (cardiopulmonary exercise testing) | Visits: Screening to Day 168
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Visits: Screening to Day 168

IPD SHARING:
Plan to Share IPD: No